CLINICAL TRIAL: NCT04594798
Title: Phase 2 Study of Polatuzumab Vedotin, Rituximab and Dose Attenuated CHP in Older Patients With DLBCL
Brief Title: A Study of Polatuzumab Vedotin, Rituximab and Dose Attenuated CHP in Older Patients With DLBCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Patrick Reagan, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULYM20030
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: DLBCL; Lymphoma, B-Cell
Keywords: polatuzumab vedotin; rituximab; cyclophosphamide; doxorubicin; prednisone; R-miniCHP; DLBCL; Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Polatuzumab Vedotin and R-CHOP (Experimental): The dose of polatuzumab vedotin for each patient will be 1.8 mg/kg (IV for 21 days)
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Polatuzumab vedotin — IV 1.8 mg/kg per cycle
Drug: Rituximab — IV 375 mg/m2 per cycle
Drug: Cyclophosphamide — IV 400 mg/m2 per cycle
Drug: Doxorubicin — IV 25 mg/m2 per cycle
Drug: Prednisone — PO 40 mg/m2 per cycle

SUMMARY:
The purpose of this study is to test the effectiveness and safety of polatuzumab vedotin in combination with R-miniCHP in patients 75 years and older with DLBCL.

DETAILED DESCRIPTION:
In this study, the investigator would like to better understand the efficacy and safety of the addition of polatuzumab vedotin to therapy with rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone (R-CHOP) and dose attenuated R-CHOP in patients who are aged 75 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-specific procedure not part of routine medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care. Subjects must be able to understand and be willing to sign the written informed consent form.
* Men and women aged greater than or equal to 75 years of age
* ECOG performance status of 0-3
* Histologically-confirmed DLBCL, NOS, NOS, high grade B-cell lymphoma with MYC, BCL2 and/or BCL6 rearrangements, high grade B-cell lymphoma, NOS, and grade 3b follicular lymphoma by 2016 WHO classification by site hematopathologist

  * Histologic transformation (HT) will be included on the study. This must be confirmed with a biopsy. Patients with HT may have received prior treatment for indolent lymphoma including chemoimmunotherapy, but must not have received an anthracycline-containing regimen in the past. Patients with Richter's transformation will be eligible.
  * Composite and discordant lymphomas containing both indolent and large cell features will be included
* Has received no prior therapy for aggressive B-cell lymphoma or HT with the following exceptions:

  * A course of corticosteroids given for lymphoma related symptoms.
  * A course of cyclophosphamide or vincristine with or without steroids given for lymphoma related symptoms.
  * One cycle of anthracycline containing chemotherapy such as R-CHOP or R-miniCHOP given urgently for aggressive disease.

Patient is not felt to be a candidate for standard dose R-CHOP due to age or comorbidities, per the site investigator.

* Ejection fraction of ≥ 45% on echocardiogram or MUGA
* Patient has a platelet count of ≥75,000/μL within 14 days before enrollment unless inadequate function is due to bone marrow infiltration with aggressive B-cell lymphoma
* Patient has an absolute neutrophil count of ≥1,500/ μL within 14 days before enrollment unless inadequate function is due to bone marrow infiltration with aggressive B-cell lymphoma
* Patient has a calculated or measured creatinine clearance of >30 mL/minute within 14 days before enrollment.
* Total bilirubin must be less than 1.5 times the upper limit of normal (ULN) unless the elevation is known to be due to Gilbert syndrome or hepatic involvement with aggressive B-cell lymphoma in which case it can be ≤ 3.0 times the ULN.
* ALT or AST must be ≤ 2.5 times the ULN.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 5 months after the last dose of polatuzumab vedotin to avoid exposing the embryo or fetus for the duration of the pregnancy. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. Male patients considering preservation of fertility should bank sperm before study treatment.

Exclusion Criteria:

* History of, or clinically apparent central nervous system (CNS) lymphoma
* Primary mediastinal B-cell lymphoma or EBV positive DLBCL
* Patient is receiving peritoneal dialysis or hemodialysis
* Patient has > Grade 1 peripheral neuropathy.
* New York Heart Association class III heart failure or EF <45%
* Patient has received other investigational drugs with 14 days before enrollment
* Prior exposure to anthracycline except for one cycle of therapy given urgently for lymphoma.
* Patient has concomitant active malignancy that the treating physician or PI feels may interfere with the ability to measure the primary or secondary outcomes

  * Patients with stage 1 cancers are eligible after definitive treatment.
  * Patients with low grade prostate cancer who are managed with observation are eligible.
  * Patients with other malignancies that have been treated with curative intent will be included if they are in documented remission without treatment for ≥ 3 years prior to enrollment.
* Patient is known to be HIV positive (test result not required for enrollment).
* Patient has active hepatitis B with a positive surface antigen or viral load. Carriers of hepatitis B virus should be closely monitored for clinical and laboratory signs of active HBV infection and for signs of hepatitis throughout study participation according to national and local guidelines. Those at high risk of reactivation should be placed on appropriate antiviral therapy as per national guidelines.
* History of solid organ transplantation, or post-transplant lymphoproliferative disorder
* Patient has history of allogeneic stem cell transplantation.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Any clinically significant abnormality in screening blood chemistry, hematology, or urinalysis results that, in the judgment of the investigator, would impede adequate evaluation of adverse

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Measure of time from study enrollment until progression.

SECONDARY OUTCOMES:
Overall Survival | From date of enrollment until date of death from any cause up to 24 months
  Measure of time from study enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Reagan, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States